CLINICAL TRIAL: NCT00005807
Title: A Phase I Scientific Exploratory Study of Epothilone B Analog in Patients With Solid Tumors and Gynecological Malignancies
Brief Title: Treating Patients With Advanced Solid Tumors, Breast Cancer or Recurrent Ovarian Cancer
Acronym: BMS-247550
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067800; AECM-9911378; NCI-98; NYU-0006
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Ovarian Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; unspecified adult solid tumor, protocol specific; ovarian stromal cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Breast Neoplasms, Male | interventions — ixabepilone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treated Participants (Experimental): dose escalation treatment
  Interventions: Drug: BMS-247550

INTERVENTIONS:
Drug: BMS-247550 — anticancer agent for the treatment of patients with malignant tumors.
  Other Names: epothilone derivative

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of BMS-247550 in treating patients who have metastatic, recurrent, or locally advanced, ovarian cancer, breast cancer, or metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, recommended phase II dose, and associated toxic effects of BMS-247550 in patients with advanced solid tumors.
* Determine the pharmacokinetic and pharmacodynamic relationship of this treatment regimen in these patients.
* Assess the extent of microtubule bundle and mitotic aster formation and cell cycle kinetics in peripheral blood mononuclear cells in these patients treated with this regimen.
* Determine any evidence of antitumor activity of this treatment regimen in these patients.
* Evaluate the relationship between tumor response and the occurrence of mutation in the class 1 isotype of B-tubulin and B-tubulin isotype distribution in patients with advanced or recurrent solid tumors, ovarian cancer, or breast cancer treated with this regimen.
* Investigate Multi-Drug Resistance Gene (MDR1), Multidrug Resistance-associated Protein (MRP) Gene, and canalicular multispecific organic anion transporter 1(cMOAT) messenger ribonucleic acid (mRNA) and protein expression as prognosticators of tumor response in these patients treated with this regimen.
* Determine the relationship between stathmin expression and phosphorylation status as a function of response in these patients treated with this regimen.
* Correlate the expression of proapoptotic (p53, bax, bad, and bid) and antiapoptotic (survivin, inhibitors of apoptotic proteins, bcl-2, and bcl-x) proteins in tumor samples and/or ascites with response and clinical outcome in these patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

* Part I: Patients with advanced solid tumors receive BMS-247550 IV over 1 hour every 3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Part II: Patients with ovarian, breast, or other cancer receive BMS-247550 as in the part I portion of the study at the MTD. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 2 months.

PROJECTED ACCRUAL: Approximately 42-66 patients will be accrued for this study within 12-16 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable solid malignancy for which no standard or curative therapies exist or are no longer effective
* Metastatic, recurrent, or locally advanced breast, ovarian, or other cancer
* Hemoglobin at least 9.0 g/dL
* WBC at least 3,000/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin normal
* AST/ALT no greater than 3 times upper limit of normal
* Gilbert's syndrome allowed
* Creatinine no greater than 2 mg/dL

Exclusion Criteria:

* symptomatic congestive heart failure
* unstable angina pectoris
* cardiac arrhythmia
* grade 2 or greater clinical neuropathy
* prior allergy or hypersensitivity reaction (grade 2 or greater) to prior paclitaxel or other therapy containing Cremophor EL
* allergy or intolerance to steroids, diphenhydramine, cimetidine, or ranitidine
* uncontrolled concurrent illness
* active infection
* pregnant or nursing
* other concurrent anticancer therapies or commercial agents
* other concurrent investigational agents
* other concurrent highly active antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-07 (Actual); Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health; Sridhar Mani, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York

REFERENCES:
- [Result] McDaid HM, Mani S, Shen HJ, Muggia F, Sonnichsen D, Horwitz SB. Validation of the pharmacodynamics of BMS-247550, an analogue of epothilone B, during a phase I clinical study. Clin Cancer Res. 2002 Jul;8(7):2035-43. PMID 12114401